CLINICAL TRIAL: NCT05086835
Title: A Mobile Executive Functioning Intervention for Momentary Craving in Opioid Use Disorders
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study ended prematurely due to PI departing institution for another position.
Sponsor: Mclean Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Andrew D. Peckham, Instructor in Psychology, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020P004112; 1K23DA051406-01A1 (NIH)
Record Dates: First submitted 2021-10-01; First posted 2021-10-21 (Actual); Results first posted 2022-06-10 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-05

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Working Memory App (Active Intervention) (Experimental): A visual-spatial app-based working memory intervention.
  Interventions: Other: Working Memory Task
- Visual Search App (Control Condition) (Active Comparator): An app-based visual search task to be used as a control condition.
  Interventions: Other: Visual Search Task

INTERVENTIONS:
Other: Working Memory Task — A smartphone-based visual-spatial working memory task that will be optimized in the Stage 1A phase of this study.
  Arms: Working Memory App (Active Intervention)
Other: Visual Search Task — A smartphone-based visual search task that will be optimized in the Stage 1A phase of this study.
  Arms: Visual Search App (Control Condition)

SUMMARY:
Even when treated with methadone or buprenorphine maintenance, many people with opioid use disorder (OUD) continue to experience craving. Among both users of heroin and users of prescription opioids, mounting evidence shows that craving predicts return to use and undermines existing treatments for OUD, thus, the development of new interventions to reduce craving is a priority for addressing the opioid crisis (NIH HEAL Initiative Research Plan, 2019). Deficits in executive functioning, particularly working memory, are a central mechanism that undermines the ability to inhibit craving. Laboratory studies in non-clinical samples show that engaging in working memory tasks before or during a craving induction increases the ability to resist craving.

This suggests that people with OUD may benefit from engaging in working memory tasks at the specific moment when craving occurs. Although previous research shows that working memory "training" does not improve clinical outcomes in OUD, these studies have not delivered training at the moment that craving actually occurs in daily life. Thus, engaging in working memory tasks at the moment that craving occurs could presumably help individuals with OUD to manage this persistent symptom, but this has not been tested.

Further, studies using Ecological Momentary Assessment (EMA) methods show that people with OUD can accurately track moment-to-moment fluctuations in craving in their daily lives, suggesting that it may be feasible to deliver interventions for craving in the moment when craving is reported. This study will test the efficacy of embedding a mobile cognitive intervention into an EMA design in people with OUD. Using the NIH Stage Model of Intervention Development, Stage 1A of this project will optimize a working memory intervention based on iterative feedback from a sample of people with OUD (n = 20), in preparation for a Stage 1B trial using a randomized design. In this trial, participants with OUDs (n = 60) will complete a two-week EMA study in which they complete smartphone-based assessments of craving five times daily. When craving is reported, a mobile application containing the working memory intervention will activate. Half of the participants will complete the intervention, while half will complete a control task. At the conclusion of the trial, participants will be granted unrestricted access to the intervention during a feasibility phase. Outcomes include change in momentary craving, change in working memory performance, and feasibility and acceptability, including use of the intervention during follow-up. Substance use will also be assessed. This project supports the applicant's goal of leveraging cognitive mechanisms to conduct treatment development research for OUD. The applicant will receive training in the etiology and treatment of OUD, craving, mobile intervention development and human-centered design of interventions, and analysis of intensive longitudinal data. With its emphasis on modifying cognitive processes at the moment of craving, using mobile devices in patients' daily lives, this project has the potential to reveal new pathways for addressing a significant predictor of relapse in OUD.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Currently receiving opioid use disorder treatment at McLean Hospital
* Primary diagnosis of opioid use disorder
* Currently prescribed medication treatment (agonist/partial agonist or antagonist) for opioid use disorder (*Note: does not apply to Stage 1A participants).
* Own a smartphone with a touchscreen and a current data plan

Exclusion Criteria:

* Acute suicidal ideation
* Acute psychosis
* Diagnosis of a neurological disorder
* History of stroke
* Diagnosis of a brain disease affecting cognitive function (e.g., tumor)
* Score of less than 26 on the Montreal Cognitive Assessment (MoCA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: By design, participants enrolled in the Stage 1A Intervention Development arm were enrolled prior to the primary clinical trial, and no data on primary study outcomes were collected during this initial treatment development phase.
Groups:
- Stage 1A Intervention Development: Adults receiving treatments for OUD. No randomization, and no intervention administered.
Period: Overall Study
Arm/Group | Stage 1A Intervention Development
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline participants in this phase did not enter into either of the study's intervention arms; by design, these participants provided feedback about the Stage 1B clinical trial design.
Groups:
- Stage 1A Intervention Development: Using the NIH Stage Model of Intervention Development, this study will consist of a non-randomized Stage 1A project designed to gather feedback from adults receiving treatments for OUD. This feedback will help our research team finalize a working memory intervention in preparation for a future Stage 1B trial using a randomized design.
Arm/Group | Stage 1A Intervention Development
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 10
Modified Credibility and Expectancy Questionnaire [Mean (Standard Deviation); unit: units on a scale] — A Modified version of the Credibility and Expectancy Scale (Devilly et al., 2000). This self-report questionnaire was used to assess participant's perceptions about the helpfulness and expected benefit of the possible study interventions to be used in the clinical trial.
  Perceived Helpfulness questions were rated on a 1-9 scale. Higher scores indicate greater perceived helpfulness.
  Perceived benefit questions were rated on a 0-100 scale. Higher scores indicate greater perceived benefit.
  units on a scale
    Perceived helpfulness of Tetris Working Memory Task | 6.5 (2.4)
    Perceived benefit (expected improvement in craving) for Working Memory Tetris Task | 65.5 (28.2)
    Perceived helpfulness of control visual search task | 4.4 (2.7)
    Perceived benefit (expected improvement in craving) for control visual search task | 41.7 (28.9)
Daily Questions Survey [Count of Participants; unit: Participants] — "Imagine that you are in a study where you are asked to use your smartphone to answer some survey questions every day. Thinking about the craving questions above, how many times per day would you be willing to answer this type of question?"
  Participants
    3 times a day (e.g., once in the morning, at midday, and in the afternoon) | 7
    Once a day | 2
    5 times a day (e.g., about every 2-3 hours) | 1

OUTCOME MEASURES:

1. Primary Outcome: Modified Craving Scale
Description: A single-item craving measure adapted from the 3-Item Craving Scale (Weiss et al., 2003).
Time Frame: Change from pre-task to immediately post-task
Population: This study was terminated prior to enrolling participants in either of the clinical trial study arms, so no outcome data were collected. Baseline data on the 10 participants who entered the Stage 1A study (designed to help inform the development of the clinical trial) are provided in the Baseline Characteristics section.
Arm/Group | Working Memory App (Active Intervention) | Visual Search App (Control Condition)
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Dot Matrix Working Memory Task
Description: A computerized version of a visual-spatial working memory task.
Time Frame: Change from baseline to post-trial (at 2 weeks)
Population: as for outcome 1
Arm/Group | Working Memory App (Active Intervention) | Visual Search App (Control Condition)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 hour
Description: This study was terminated prior to enrolling participants in either of the clinical trial study arms, so the number of participants at risk for Serious Adverse Events in the planned clinical trial is zero. All-cause mortality, and Other Adverse Events is 0 for both study arms.
  In addition, there were no Serious Adverse Events nor Other Adverse Events recorded in the participants enrolled in the Stage 1A phase (n = 10 participants total).
Arm/Group | Working Memory App (Active Intervention) | Visual Search App (Control Condition) | Stage 1A Intervention Development
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/10
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/10

LIMITATIONS AND CAVEATS:
This study was terminated prior to enrolling participants in either of the clinical trial study arms, so no outcome data were collected. Baseline data on the 10 participants who entered the Stage 1A study (designed to help inform the development of the clinical trial) are provided in the Baseline Characteristics section.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-09): https://cdn.clinicaltrials.gov/large-docs/35/NCT05086835/Prot_SAP_000.pdf